CLINICAL TRIAL: NCT05359536
Title: Impact of an Early Childhood Educator e-Learning Course in Physical Activity and Sedentary Behaviour on Young Children's Movement Behaviours in Childcare: The TEACH-Preschooler Study
Brief Title: Training Early Childhood Educators to Increase Children's Physical Activity: The TEACH-Preschooler Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R4368A35
Record Dates: First submitted 2022-04-22; First posted 2022-05-04 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Physical Activity
Keywords: Physical activity; Fundamental movement skills; E-learning; Preschool
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- E-learning Intervention (Experimental): Early career educators in the intervention condition will be asked to complete a 5-hour e-learning course over a two week timeframe. The four module e-learning course was developed using the Delphi technique and covers physical activity and sedentary guidelines, physical activity and sedentary behaviours in the childcare environment, how to promote physical activity and reduce sedentary behaviours in young children, and a resource library.
  Interventions: Behavioral: Training Early Childhood educators in PA
- Usual Practice Control (No Intervention): Early career educators in the control condition will be asked to continue with their usual practices. They will be invited to complete the e-learning course after the study period.

INTERVENTIONS:
Behavioral: Training Early Childhood educators in PA — The four module e-learning course was developed using the Delphi technique and covers physical activity and sedentary guidelines, physical activity and sedentary behaviours in the childcare environment, how to promote physical activity and reduce sedentary behaviours in young children, and a resource library.
  Arms: E-learning Intervention

SUMMARY:
This study aims to determine the effect of delivering a physical activity e-learning course to early childhood educators on young children's physical activity and sedentary behaviour while at childcare. It is hypothesized that levels of physical activity will increase and levels of sedentary behaviours will decrease during time spent in childcare in a sample of children who attend early childcare centres where early childhood educators have completed the physical activity e-learning course compared to children in centres where early childhood educators are randomized to not receive the intervention. Differences in changes in several secondary outcomes including fundamental movement skills, parent's perceptions of children's fundamental movement skills, children's cognitive development, emotional symptoms, conduct problems, hyperactivity/inattention, peer relationship problems and prosocial behaviours will also be examined.

DETAILED DESCRIPTION:
In this cluster randomized controlled trials, early childhood educators from childcare centres in London, Ontario, Canada will be randomized to complete a 4 module e-learning course with content on physical activity and sedentary guidelines, physical activity and sedentary behaviours in the childcare environment, how to promote physical activity and reduce sedentary behaviours in young children, and a resource library, or to continue with their usual practices. Early childhood educators randomized to the intervention group will be asked to complete this course over a 2-week intervention period.

In both the intervention and control groups, preschoolers physical activity and sedentary behaviours will be measured at baseline, post-intervention (2-weeks) and 3-months follow-up using Actigraph GT3X+ accelerometers. Preschoolers will also complete tasks at baseline and 3-month follow-up to measure their cognitive development, and a subgroup of randomly selected children from each group will complete the Tests of Gross Motor Development - Third Edition to assess their fundamental movement skill proficiency at baseline and follow-up. Parents of children in both groups will complete a questionnaire to measure their perception of their children's proficiency at fundamental movement skills. Parents will also be asked to report on their child's emotional symptoms, conduct problems, hyperactivity/inattention, peer relationship problems and prosocial behaviours by completing the Strength and Difficulties Questionnaire

ELIGIBILITY:
Inclusion Criteria:

Childcare Centres:

* Located in London, ON, Canada
* Have at least 1 preschool classroom
* Open every weekday
* Operate for at least 8 hours on weekdays
* All early childhood educators are willing to participate in the study
* Staff are English speaking

Early Childhood Educators:

* Employed at a participating childcare centre
* English speaking

Children:

* Enrolled at a participating childcare centre
* Between the ages 2.5-5 years at baseline
* Are expected to remain at the childcare centre for the duration of the study period

Exclusion Criteria:

Childcare Centres:

* Not located in London, ON, Canada
* Do not have at least 1 preschool classroom
* Not open every weekday
* Do not operate for at least 8 hours on weekdays
* Not all early childhood educators are willing to participate in the study
* Staff do not speak English

Early Childhood Educators:

* Not employed at a participating childcare centre
* Do not speak English

Children:

* Not enrolled at a participating childcare centre
* Not between the ages 2.5-5 years at baseline
* Not expected to remain at the childcare centre for the duration of the study period

Ages: 30 Months to 60 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 145 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2023-08-28 (Actual); Study Completion 2023-08-28 (Actual)

PRIMARY OUTCOMES:
Change in children's device measured moderate-to-vigorous physical activity while at childcare measured | Baseline, post-intervention (2-weeks), and 3-months follow-up
  Assessed using ActiGraph GT3X+ accelerometers worn on each child's right hip for 5 consecutive days (Monday-Friday) while at childcare. Age-specific validated accelerometer cut-points will be used to calculate time spent in moderate-to-vigorous physical activity (i.e. >420 counts/15-second epoch). Children will be considered to have valid accelerometer data if they have at least 5 hours of accelerometer data on 2 days. Accelerometer non-wear time will be identified as any period with 20 consecutive minutes of zero counts.

SECONDARY OUTCOMES:
Change in children's device sedentary behaviours while at childcare | Baseline, post-intervention (2-weeks), and 3-months follow-up
  Assessed using ActiGraph wGT3X-BT accelerometers worn on each child's right hip for 5 consecutive days (Monday-Friday) while at childcare. Age-specific validated accelerometer cut-points will be used to calculate time spent in moderate-to-vigorous physical activity (i.e. <48 counts/15-second epoch). Children will be considered to have valid accelerometer data if they have at least 5 hours of accelerometer data on 2 days. Accelerometer non-wear time will be identified as any period with 20 consecutive minutes of zero counts.
Change in children's fundamental movement skills | Baseline and 3-months follow-up
  Assessed in a sub-sample of randomly selected children using the Test of Gross Motor Development - Third Edition. Test of Gross Motor Development - Third Edition tests six locomotor skills (run, gallop, hop, skip, jump, and slide) and 7 object control skills (two handed strike, forehand strike, dribble, catch, kick, overhand throw, and underhand throw). Each skill was assessed and scored twice on between 3-5 performance criteria where a child was given a 1 if the skill is performed correctly and a 0 if performed incorrectly. A total score between 0-100 is calculated with a higher score indicating a better outcome.
Change in parent's perceptions of fundamental movement skill proficiency | Baseline and 3-months follow-up
  Parents of children will be asked to report their perceptions of their child's fundamental movement skills. The self-reported scale will measure the same 13 fundamental movement skills measured in the Test of Gross Motor Development - Third Edition. The will rate their Childs proficiency for each skill on a scale from 1 = not that good, 2 = sort of good, 3 = pretty good and 4 = really good. Eah skill is presented with a picture of the skill being performed. The range of possible scores for this scale are 13-52, with higher scores indicating a better outcome.
Changes in scores on the Strengths and Difficulties Questionnaire | Baseline and 3-months follow-up
  Parents will report on their child's emotional symptoms, conduct problems, hyperactivity/inattention, peer relationship problems and prosocial behaviours. Each item is scored on a scale from 0 =not true, 1 =somewhat true, and 2 = certainly true, with positively worded questions being reversed scored for the emotional symptoms, conduct problems, hyperactivity/inattention, and peers relationship problem subscales. Higher scores on these four subscales indicates a worse outcome, while a higher score on the emotional symptoms subscale indicates a better outcome. Each subscale is scored on a scale from 0-10.

CONTACTS AND LOCATIONS:
Locations (1):
- Child Health and Physical Activity Lab, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Phillips SM, Bourke M, Bruijns BA, Vanderloo L, Loh A, Saravanamuttoo K, Tucker P. Associations Between Childcare Physical Activity and Sedentary Time and Early Childhood Developmental Outcomes: A Compositional and Isotemporal Substitution Analysis. Child Care Health Dev. 2024 Nov;50(6):e70011. doi: 10.1111/cch.70011. PMID 39569560